CLINICAL TRIAL: NCT00532012
Title: An Open-Label, Partially Randomized, Cross-Over, Monocentric Phase I Study Evaluating the Pharmacokinetic Profile of RhuDex® in Order to Determine Optimum Doses of Meglumine and RhuDex®
Brief Title: Phase-I Study Evaluating the Pharmacokinetic Profile of RhuDex®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MediGene (Industry)
Responsible Party: Hoda Tawfik / Clinical Trial Manager, MediGene
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CT 5001
Record Dates: First submitted 2007-09-18; First posted 2007-09-19 (Estimated); Last update posted 2008-07-16 (Estimated); Status verified 2008-07

CONDITIONS: Pharmacokinetics
Keywords: Rheumatoid Arthritis; RhuDex®; Meglumine; Oral Bioavailability
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: RhuDex®

SUMMARY:
The drug that is under investigation during this study is RhuDex® and is expected to be used as an oral treatment for rheumatoid arthritis. Normal stomach juices contain acid and previous studies have shown that this acidity reduces the solubility and therefore the absorption of RhuDex®. Administering the alkaline buffer meglumine with RhuDex® has shown to increase the solubility of RhuDex® by decreasing the stomach acidity.

The purposes of this study are to determine:

* the optimum level of meglumine which is required to achieve the best uptake of RhuDex® from the stomach into the blood
* to determine the concentration of RhuDex® in the blood in the presence of the optimum level of meglumine
* to investigate further the safety and tolerability of RhuDex®. The study will be conducted in healthy male volunteers.

DETAILED DESCRIPTION:
RhuDex® is a novel, orally bioavailable, low molecular weight modulator of co-stimulation of T lymphocytes. RhuDex® binds to the protein CD80 on the surface of antigen-presenting cells and inhibits its interaction with CD28 (but not with CTLA-4) presented by CD4+ T lymphocytes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between 18 and 60 years at the time of enrollment
* Male volunteers and their partners who are of child-bearing potential must agree to use a double-barrier method of contraception during the study and for 12 weeks after discharge
* BMI between 18.5 and 29.9 kg/m²
* Written informed consent
* Ability to comply with the requirements of the study

Exclusion Criteria:

* Acute infection at time of enrollment
* History of chronic inflammation, chronic infection, other chronic disease, autoimmune disorders (e.g. diabetes mellitus) or cancer
* Clinical significant abnormal ECG
* Clinical significant abnormal laboratory values (especially in terms of liver or renal insufficiency)
* Clinically significant physical findings
* Major surgery within the last 4 weeks prior to enrollment
* Organ allograft recipient
* Concomitant or planned treatment which would interfere with study results
* Any systemic medical treatment, including over the counter products and dietary supplements such as iodine, fluoride or vitamins, within one week before and during the study course
* Known allergy against any ingredient of the study medication or meglumine
* Participation in an investigational trial within 30 days prior to enrollment
* Systemic intake of immunosuppressive or immunomodulatory medication or vaccination within 30 days prior to enrollment and for the whole study duration
* Blood loss exceeding 450 mL (including blood donations) within 12 weeks prior to enrollment into the study
* Medical history of alcohol or drug abuse or alcohol consumption greater than 21 units per week for males. A unit of alcohol is equivalent to: half a pint of average strength beer (280 mL), a glass (125 mL) of wine or a standard measure (25 mL) of spirits, sherry or port
* A positive alcohol breath test
* A positive urine drug screen
* Regular smokers (more than 20 cigarettes or 5 cigars per day)
* Presence of hepatitis B surface antigen (HBsAG), hepatitis C antibody (HCV Ab) or HIV-1 or HIV-2 antibodies at screening

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2007-09; Primary Completion 2007-10 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Profile

SECONDARY OUTCOMES:
Safety Profile

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Freestone, MD, Principal Investigator — Syneos Health
Locations (1):
- Charles River Clinical Services Edinburgh Ltd, Edinburgh, United Kingdom